CLINICAL TRIAL: NCT01521624
Title: Comparing Effects of Metformin Plus Life Style Modification Compared With Life Style Modification Alone in Lowering Parameters of Oxidative Stress in Newly Diagnosed Type 2 Diabetes Patients
Brief Title: Metformin Effects on Oxidative Stress Parameters in Newly Diagnosed Type 2 Diabetes Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Alireza Esteghamati, Professor Alireza Esteghamati, Tehran University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 90-01-30-13350
Record Dates: First submitted 2012-01-26; First posted 2012-01-30 (Estimated); Last update posted 2012-01-31 (Estimated); Status verified 2012-01

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Case (Active Comparator): Metformin 1000 mg Daily in two divided doses plus advice for lifestyle modification
  Interventions: Drug: Metformin
- Control (No Intervention): Subjects provided only advice for lifestyle modification with no drug intervention

INTERVENTIONS:
Drug: Metformin — Metformin 1000 mg Daily in two divided doses plus advice for lifestyle modification
  Arms: Case

SUMMARY:
Oxidative stress plays a key role in the pathogenesis of diabetes complications. Chronic hyperglycemia and disturbed lipid regulation commonly seen in diabetes are the main causes of this process. Despite the critical role of oxidative stress in diabetes, most clinical trials with available antioxidants and vitamins have either failed to show any long term benefits or have produced inconsistent results (10-11). There has been growing interest in establishing the possible roles of oral hypoglycemic agents including Metformin in reduction of oxidative stress. Metformin, the most common prescribed oral medication in type 2 diabetes, lowers HbA1c around 1.5%, rarely causes hypoglycemia (compared with insulin or sulfonylureas), has relatively few contraindications, its adverse effects are generally tolerable, does not cause weight gain, is cheap, and is highly acceptable among patients. Given the long term benefits observed with metformin use, a role in modulating oxidative stress is imputable. We designed this study to evaluate the actions of metformin on oxidative stress in a group of medication-naïve newly diagnosed type 2 diabetes patients.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed type 2 diabetes patients based on American Diabetes Association criteria for diagnosis of diabetes

Exclusion Criteria:

* No history of serious chronic illnesses of heart, lung, and kidney
* No prior treatment with anti-diabetes medications for either diabetes or conditions associated with hyperglycemia
* No intake of prescribed or over-the-counter vitamins C and E in the past year; - No intake of aspirin in the past year
* No history of excessive alcohol intake in the past year

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2010-10; Primary Completion 2011-03 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Serum concentrations of various markers of oxidative stress | 12 weeks
  Serum concentrations of markers of oxidative stress (i.e. advanced glycation end products, advanced oxidation protein products, ferritin reducing ability of plasma) along with activities of antioxidant enzymes (i.e. paraoxonase1, lecithin cholesterol asyltransferase) are measured. To assess the change in inflammatory condition associated with fat tissue dysfunction (a close entity to oxidative stress) serum concentrations of fat tissue hormones (i.e. leptin, vaspin, adiponectin, visfatin)are also assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Alireza Esteghamati, M.D., Principal Investigator — Tehran University of Medical Sciences
Locations (1):
- Tehran University of Medical Sciences, Tehran, Tehran Province, Iran

REFERENCES:
- [Derived] Esteghamati A, Rezvani S, Khajeh E, Ebadi M, Nakhjavani M, Noshad S. Comparative effects of metformin and pioglitazone on YKL-40 in type 2 diabetes: a randomized clinical trial. J Endocrinol Invest. 2014 Dec;37(12):1211-8. doi: 10.1007/s40618-014-0154-x. Epub 2014 Aug 20. PMID 25138574
- [Derived] Mirmiranpour H, Mousavizadeh M, Noshad S, Ghavami M, Ebadi M, Ghasemiesfe M, Nakhjavani M, Esteghamati A. Comparative effects of pioglitazone and metformin on oxidative stress markers in newly diagnosed type 2 diabetes patients: a randomized clinical trial. J Diabetes Complications. 2013 Sep-Oct;27(5):501-7. doi: 10.1016/j.jdiacomp.2013.05.006. Epub 2013 Jul 23. PMID 23891275
- [Derived] Esteghamati A, Eskandari D, Mirmiranpour H, Noshad S, Mousavizadeh M, Hedayati M, Nakhjavani M. Effects of metformin on markers of oxidative stress and antioxidant reserve in patients with newly diagnosed type 2 diabetes: a randomized clinical trial. Clin Nutr. 2013 Apr;32(2):179-85. doi: 10.1016/j.clnu.2012.08.006. Epub 2012 Aug 21. PMID 22963881